CLINICAL TRIAL: NCT07096141
Title: Improving Emotional Wellbeing of University Students Using Culturally Adapted Dialectic Behaviour Approaches in Group Settings" (UniWELL-D): Protocol of a Feasibility and Effectiveness Study
Brief Title: Improving Emotional Wellbeing of University Students: Emotion Regulation
Acronym: UniWELL-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bogazici University (Other)
Responsible Party: Principal Investigator, Ayse Akan, Assistant Professor and Clinical Psychologist, Bogazici University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20022
Record Dates: First submitted 2025-04-14; First posted 2025-07-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Emotion Regulation
Keywords: emotion regulation; mental health; DBT; group therapy; university student mental health; culturally adapted psychotherapy
MeSH Terms: conditions — Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single-centre interventional non-blinded mixed-methods non-randomised pre-post design with a waitlist control and 6 weeks follow-up feasibility and psychotherapy effectiveness study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT Experimental Arm (Experimental): An 8-session Dialectical Behaviour Therapy informed emotional regulation group psychotherapy will be offered to the experimental group of about 40 university students who volunteered and scored above the threshold on the Difficulties in Emotion Regulation Scale (DERS-16).
  Interventions: Behavioral: DBT-informed Group Psychotherapy for Emotion Regulation
- DBT Waitlist Arm (No Intervention): DBT waitlist control

INTERVENTIONS:
Behavioral: DBT-informed Group Psychotherapy for Emotion Regulation — An 8-session Dialectical Behaviour Therapy informed emotion regulation psychotherapy group.
  Other Names: DBT; Group DBT
  Arms: DBT Experimental Arm

SUMMARY:
University students' psychological well-being is a growing public health concern. University life involves major psychological, social, and academic changes, increasing vulnerability to mental health issues. Group-based Dialectical Behaviour Therapy (DBT) has been shown to support student well-being effectively. However, interventions tailored to specific cultural and contextual needs are more likely to be helpful. Western-based therapy models may not fully align with non-Western populations, such as students in Türkiye.

In Türkiye, public mental health services are often limited to short psychiatric consultations, while therapy is typically accessed privately. University counselling centres offering free or low-cost therapy are therefore essential. Cost-effective interventions like group DBT may be especially valuable in these settings. To address this gap, culturally adapted DBT groups should be developed and evaluated for Turkish university students.

This study is part of the UniWELL Project (sister to UniWELL-C) and examines the effectiveness of DBT-informed emotion regulation groups for Turkish students. Any Bogazici University student aged 18+ is eligible. Exclusion criteria include severe mental illness, high risk of harm to self/others, or scoring below threshold on the Difficulties in Emotion Regulation Scale (DERS-16), as these students may require more individual support.

The study includes participation in an 8-session DBT-informed group. Participants are expected to benefit from free psychological support, guided reflection, and shared experiences with peers. The research will also contribute to the evidence base for culturally adapted interventions.

There are some risks: participants may feel overwhelmed during the sessions or while completing questionnaires. If so, support will be provided by a clinical psychology master's student and/or the group facilitator, under supervision of an experienced clinical psychologist. If a participant's risk increases, they will be referred to psychiatric services. An emergency contact will be requested to ensure safety if needed.

The study will take place at Bogazici University through the Translational Clinical Psychology Lab, in collaboration with BUREM. It is expected to run for at least one year, possibly extending up to three years. The study is partially funded by the Bogazici Scientific Research Projects Unit (20022). Dr Ayse Akan (t-clinpsylab@bogazici.edu.tr) is the study lead and main contact.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a Bogazici University student.
2. Must be 18 years or older.
3. Must score above the threshold on the Difficulties in Emotion Regulation Scale (DERS-16).

Exclusion Criteria:

1. Not Bogazici University student.
2. Has serious and severe mental illness.
3. High risk of self-harm/harm to others.
4. Scoring below the threshold of on the Difficulties in Emotion Regulation Scale (DERS-16).
5. Younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS-16) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion intervention
  Difficulties in Emotion Regulation Scale (DERS-16) is a questionnaire that measures different aspects of difficulties in emotion, including emotional awareness, clarity, acceptance, impulse control, and goal-directed behavior during emotional distress. Each item is scored on a 5-point Likert scale, from 1 (almost never) to 5 (almost always), resulting in a total score range of 16 to 80. Higher scores indicate greater difficulties in emotion regulation.

SECONDARY OUTCOMES:
Borderline Evaluation of Severity Over Times (BEST) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion intervention
  The Borderline Evaluation of Severity Over Times (BEST) is a tool that measures the severity and progression of thoughts, feelings, and behaviors that are typical of Borderline Personality Disorder. Each item is rated on a 5-point Likert scale, where 1 indicates none/rarely and 5 indicates almost always, resulting in a total score range between 12 and 72. Higher scores indicate more severe symptoms. The scale also provides information about positive behaviors separately.
Depression Anxiety and Stress Scale (DASS-42) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion of the intervention
  Depression Anxiety Stress Scale (DASS-42) is a questionnaire that measures the negative emotional states depression, anxiety and stress. Each subscale is scored separately. Each item is rated on a 4-point Likert scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Scores for each subscale range from 0 to 42, and the combined total scale ranges from 0 to 126. Higher scores indicate more severity. The severity is categorized into "normal", "mild", "moderate", "severe", and "extremely severe".
Generalised Anxiety Disorder-7 (GAD7) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion of the intervention
  The Generalised Anxiety Disorder - 7 Scale (GAD7) is a questionnaire used to screen for Generalised Anxiety Disorder and assess the severity of anxiety symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 21. Higher scores indicate more severity. The severity is categorized into "minimal", "mild", "moderate", and "severe".
Patient Health Questionnaire (PHQ9) | Baseline, immediately after the intervention, and follow-up 6 weeks after the completion of the intervention
  The Patient Health Questionnaire (PHQ9) is a scale used for assessing the presence and the severity of depression. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), resulting in a total score that ranges from 0 to 27. Higher scores indicate more severity of depressive symptoms. The severity is categorized into "minimal", "mild", "moderate", "moderately severe" and "severe".
Outcome Rating Scale (ORS) | From enrollment to the end of treatment at 8 weeks
  Outcome Rating Scale (ORS) is a brief 4-item scale used for assessing the members' overall functioning in key areas: individual well-being, interpersonal relationships, social role, and overall well-being. Each item is rated on a visual analog scale from 0 to 10, resulting in a total score between 0 and 40. Higher scores indicate better overall functioning and well-being.
Qualitative data | Up to 12 weeks following the completion of the intervention
  Participants who completed their groups will also be invited to attend a semi-structured interview for in-depth qualitative feedback when they finish the intervention. Below are the sample questions to be asked to the participants:
  1. Could you tell us a little about the process (your mental health difficulties) that led you to apply to this group?
  2. Were you satisfied with the group?
  3. Which parts of the group were useful to you?
  4. Which parts of the group need to change (what you didn't like)?
  5. How was your relationship with the therapist and assistants?
  6. How was your relationship with the other participants of the group?
  7. What was the most important thing you learned from the group?
  8. Are there any other things that stood out to you?
  9. Would you recommend this group to other students with similar problems?
  10. Do you think this group should be an ongoing service provided by the university?

OTHER OUTCOMES:
Group Session Rating Scale (GSRS) | From enrollment to the end of treatment at 8 weeks
  Group Session Rating Scale (GSRS) is a brief 4-item scale used for assessing the members' evaluation of each session regarding the therapeutic relationship, goals and topics, approach or method, and overall experience. Each item is rated on a visual analog scale from 0 to 10, resulting in a total score between 0 and 40. Higher scores indicate more satisfaction with the group session.
Feedback Form | Immediately after the intervention
  The client feedback form is a 4-point self-report scale with a free-text box for additional comments. It is used to gather information about participants' experiences with the group facilitator and the intervention. The form includes questions about the therapeutic process, the structure of the sessions, the therapist's approach, and whether the support was helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Akan, DClinPsych, Principal Investigator — Bogazici University
Locations (2):
- Turkey (Türkiye) (2):
  - Bogazici University Student Guidance and Psychological Counselling Centre (BUREM), Istanbul
  - Translational Clinical Psychology Lab, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
The anonymised quantitative data will be kept securely on a password protected drive for 10 years and will be shared with peer-reviewers if requested, while the qualitative interview transcripts will also be kept securely on a password protected drive but they will not be shared with peer-reviewers (will be only open to the research team) until it is deleted after 10 years. Some of the research team may use these data in secondary analysis projects.
Time Frame: The data supporting this study's findings will be available from the corresponding author upon reasonable request, starting immediately after publication. Data will be maintained and available for 10 years after the last data collection.
Access Criteria: Being a peer-reviewer / researcher.